CLINICAL TRIAL: NCT01568333
Title: A Multi-center Study of Low-dose Decitabine for the Treatment of Immune Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Qingdao University (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITP-Low-dose Decitabine; 81270578 (Other Grant/Funding Number: Natural Science Foundation of China)
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Immune Thrombocytopenia
Keywords: Decitabine; Immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine (Experimental): Decitabine 3.5mg/m2，ivdrip，qd x 3d, every four weeks for one cycle. It will be given three cycles.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine 3.5mg/m2，ivdrip，qd x 3d, every four weeks for one cycle. It will be given three cycles.

SUMMARY:
Decitabine has been reported to have a clinically significant, often long lasting effect on the platelet count in myelodysplastic syndromes(MDS). It is also reported that decitabine could increase platelet counts by enhancing megakaryocyte maturation and platelet release. Immune thrombocytopenia(ITP) is known as an immune-mediated acquired disease characterized by transient or persistent decrease of the platelet count. However, refractory ITP is lacking of effective treatments and the efficacy of decitabine in ITP remains poorly understood. Data from this study may provide some idea of decitabine in the treatment of ITP.

DETAILED DESCRIPTION:
The investigators are undertaking a multicenter, single-arm study of primary ITP adult patients from 9 medical centers in China. All the participants are selected to receive low-dose of decitabine treatment (given intravenously at a dose of 3.5mg/m2 for 3 days per cycle for 3 cycles). Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with the diagnosis of ITP according to the International Working Group (IWG) guidelines
* failure to splenectomy or at least four standard ITP-specific treatments, but not necessarily undergone splenectomye
* baseline peripheral platelet count less than 30,000/uL or the presence of bleeding symptoms
* need of treatment(s) (including, but not limited to, low dose of corticosteroids) to minimize the risk of clinically significant bleeding. Need of on-demand or

Exclusion Criteria:

* secondary ITP
* pregnancy
* hypertension
* cardiovascular disease
* diabetes
* liver and kidney function impairment
* HCV, HIV, HBsAg seropositive status
* patients with systemic lupus erythematosus and/or antiphospholipid syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Platelet count | the third month after the first dose of decitabine
  plate level at the third month after the first dose of decitabine

SECONDARY OUTCOMES:
Bleeding score | at enrollment and the third month after the first dose of decitabine
  the assessment of bleeding scores at enrollment and at the third month after the first dose of decitabine

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Shandong University Qilu hospital, Jinan, Shandong, China

REFERENCES:
- [Background] van den Bosch J, Lubbert M, Verhoef G, Wijermans PW. The effects of 5-aza-2'-deoxycytidine (Decitabine) on the platelet count in patients with intermediate and high-risk myelodysplastic syndromes. Leuk Res. 2004 Aug;28(8):785-90. doi: 10.1016/j.leukres.2003.11.016. PMID 15203276
- [Background] Wang J, Yi Z, Wang S, Li Z. The effect of decitabine on megakaryocyte maturation and platelet release. Thromb Haemost. 2011 Aug;106(2):337-43. doi: 10.1160/TH10-11-0744. Epub 2011 Jun 28. PMID 21713321
- [Derived] Zhou H, Qin P, Liu Q, Yuan C, Hao Y, Zhang H, Wang Z, Ran X, Chu X, Yu W, Wang X, Hou Y, Peng J, Hou M. A prospective, multicenter study of low dose decitabine in adult patients with refractory immune thrombocytopenia. Am J Hematol. 2019 Dec;94(12):1374-1381. doi: 10.1002/ajh.25646. Epub 2019 Oct 17. PMID 31591739